CLINICAL TRIAL: NCT00066274
Title: Randomized Phase II Study Evaluating Three Chemotherapies: [Irinotecan + Oxaliplatin (Irinox)], [Irinotecan + LV5FU2] and [Oxaliplatin + LV5FU2] as First Intention Treatment in Subjects With Metastatic Colorectal Cancer
Brief Title: Comparison of Combination Chemotherapy Regimens in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: Accord 08; FRE-FNCLCC-ACCORD-08/0103; EU-20233
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving the drugs in different combinations may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying combination chemotherapy containing irinotecan and oxaliplatin to see how well it works compared to two standard combination chemotherapy regimens in treating patients with unresectable metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy, in terms of response rate (partial response and complete response), of irinotecan and oxaliplatin vs irinotecan, fluorouracil, and leucovorin calcium vs oxaliplatin, fluorouracil, and leucovorin calcium in patients with metastatic colorectal cancer.
* Compare the progression-free survival of patients treated with these regimens.
* Compare the tolerability of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive irinotecan IV over 90 minutes and oxaliplatin IV over 2 hours on day 1.
* Arm II: Patients receive irinotecan IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours on days 1-2.
* Arm III: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours on days 1-2.

In all arms, treatment repeats every 2 weeks for 26 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 3 months for 1 year.

Patients are followed at 2 months.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal carcinoma

  * Metastatic disease
* Not amenable to surgery
* Unidimensionally measurable disease
* No bone metastases
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* WHO 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than 1.25 times upper limit of normal (ULN) (1.5 times ULN if hepatic metastases are present)
* SGPT and SGOT no greater than 3 times ULN (5 times ULN if hepatic metastases are present)

Renal

* Creatinine no greater than 1.25 times ULN

Cardiac

* No concurrent cardiac abnormalities that would preclude study therapy

Pulmonary

* No concurrent pulmonary abnormalities that would preclude study therapy

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No chronic enteropathy
* No other prior cancer within the past 5 years except carcinoma in situ of the cervix or curatively treated basal cell skin cancer
* No concurrent severe uncontrolled infection
* No obstruction or partial obstruction that would interfere with study therapy
* No psychological, social, familial, or geographical situation that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer biological response modifiers

Chemotherapy

* No prior chemotherapy (except adjuvant chemotherapy completed more than 6 months ago)
* No prior irinotecan
* No prior oxaliplatin
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent anticancer hormonal therapy

Radiotherapy

* At least 4 weeks since prior pelvic radiotherapy
* No prior abdominopelvic radiotherapy

Surgery

* At least 4 weeks since prior surgery
* No prior extensive intestinal resection (i.e., more than 1 prior hemicolectomy or extensive resection of the small intestines)

Other

* No other concurrent experimental medication
* No other concurrent anticancer therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-07-23 (Actual); Primary Completion 2005-11-04 (Actual); Study Completion 2007-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves Becouarn, MD, Study Chair — Institut Bergonié
Locations (17):
- France (17):
  - Centre Hospitalier de L' Agglomeration Montargoise, Amilly
  - Pole Sante Sarthe et Loir Hopital Pierre Daguet, Angers
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Clinique Sainte-Marguerite, Hyères
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Polyclinique Francheville, Périgueux
  - Centre Eugene Marquis, Rennes
  - CHG Roanne, Roanne
  - Centre Hospitalier de Rodez, Rodez
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier Regional Metz Thionville, Thionville
  - Centre Hospitalier General Lucien Hussel, Vienne

REFERENCES:
- [Result] Becouarn Y, Senesse P, Thezenas S, Boucher E, Adenis A, Cany L, Jacob JH, Cvitkovic F, Montoto-Grillot C, Ychou M; Digestive Group of the Federation Nationale des Centres de Lutte Contre le Cancer. A randomized phase II trial evaluating safety and efficacy of an experimental chemotherapy regimen (irinotecan + oxaliplatin, IRINOX) and two standard arms (LV5 FU2 + irinotecan or LV5 FU2 + oxaliplatin) in first-line metastatic colorectal cancer: a study of the Digestive Group of the Federation Nationale des Centres de Lutte Contre le Cancer. Ann Oncol. 2007 Dec;18(12):2000-5. doi: 10.1093/annonc/mdm379. Epub 2007 Sep 4. PMID 17785765